CLINICAL TRIAL: NCT04746222
Title: Oral Capsule-administered Faecal Microbiota Transplantation for Intestinal Carbapenemase-producing Enterobacteriaceae Decolonization
Brief Title: Oral Capsule Faecal Microbiota Transplantation for CPE Decolonization
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSAINV18nov-006
Record Dates: First submitted 2021-02-07; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomised controlled trial to evaluate the clinical efficacy of oral capsule administered FMT for CPE-intestinal decolonisation compared with placebo (1:1)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects will be randomised to either FMT-capsules or placebo (subject and investigator-blinded) immediately prior to capsule administration. Subjects who are randomised to FMT by capsule will receive 30 FMT-containing capsules under direct-observed therapy. Subjects who are randomised to placebo capsules will receive 30 placebo capsules under direct-observed therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Single dose of 30 oral capsules containing FMT from a stool bank
  Interventions: Biological: Oral capsule faecal microbiota transplantation
- Placebo (Placebo Comparator): Single dose of 30 oral placebo capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Oral capsule faecal microbiota transplantation — Single dose of 30 oral capsules containing healthy donor stool from a stool bank
  Arms: Treatment
Other: Placebo — Single dose of 30 oral placebo capsules
  Arms: Placebo

SUMMARY:
Double-blinded, randomised controlled trial to evaluate the clinical efficacy of a single dose of oral capsule-administered faecal microbiota transplantation (FMT) for carbapenemase-producing Enterobacteriaceae (CPE) intestinal decolonisation compared with placebo. Primary outcome is the proportion of patients successfully decolonised of CPE intestinal carriage at 12 weeks after FMT treatment compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Admitted as inpatient at the study site at the time of screening.
* Aged ≥21 years at the time of screening.
* Sufficiently ambulant to return for outpatient clinic study visit.
* Detection of CPE (result reported by clinical microbiology laboratory).
* Ability to provide informed consent.
* Females of childbearing potential who are sexually active with a non-sterilised male partner must agree to use at least one method of effective contraception for the duration of the trial.
* Colonisation of the gastrointestinal tract with CPE, confirmed by at least one positive rectal swab taken ≤7 days before randomisation (direct PCR testing using Xpert Carba-R, performed by study team independent of the hospital screening protocol).
* Ability to swallow "safety test" capsule (one test capsule given during pre-randomisation evaluation).
* Antibiotics ceased for at least 48 hours before pre-randomisation evaluation.
* Negative urine pregnancy test for pre-menopausal women taken ≤7 days before randomisation

Exclusion Criteria:

* Presence of acute diarrhoeal illness (e.g. gastroenteritis, C. difficile colitis) or chronic diarrhoeal illness (e.g. irritable bowel syndrome or inflammatory bowel disease, unless they are in remission for at least 3 months prior to enrolment).
* Current use or planned use of an investigational drug within 3 months of enrolment.
* Presence of significant immunosuppression, including but not limited to: use of monoclonal antibody, use of prolonged steroids equivalent to prednisolone dose of ≥20mg/day for ≥28 days, solid organ transplantation, bone marrow transplantation, HIV infection with CD4 count of ≤200, bone marrow transplant, ongoing chemotherapy or radiation therapy, and congenital immunodeficiency.
* Oropharyngeal dysphagia, significant oesophageal dysphagia, or other inability to swallow.
* History of surgery altering gastrointestinal anatomy (e.g. colostomy, colectomy).
* Ileus or small bowel obstruction.
* Risk of aspiration.
* History of gastroparesis.
* Severe food allergy (anaphylaxis or anaphylactoid reaction).
* Adverse event attributable to previous FMT.
* Those who are pregnant or plan to be pregnant within 3 months of enrolment.
* Those who are breastfeeding or plan to breastfeed during the trial.
* Life expectancy <3 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients successfully decolonised of CPE intestinal carriage at 12 weeks. | 12 weeks
  Decolonisation is determined by the following test outcomes:
  i. Negative PCR result (CP genes undetected) for rectal swab sample subjected to direct PCR (Xpert Carba-R) ii. Negative PCR result (CP genes undetected) for rectal swab sample subjected to culture on ChromID CARBA SMART media followed by PCR for suspected CPE colonies (Xpert Carba-R) iii. Negative PCR result (CP genes undetected) for stool sample subjected to direct PCR (Xpert Carba-R) iv. Negative PCR result (CP genes undetected) for stool sample subjected to culture on ChromID CARBA SMART media followed by PCR for suspected CPE colonies (Xpert Carba-R)
  At least two of the four tests must be evaluable (clear positive or negative result obtained). Subject not meeting these criteria will be considered not-decolonised.
  If any one of the PCR results are positive, the subject is considered not-decolonised.

SECONDARY OUTCOMES:
Proportion of patients successfully decolonised of CPE intestinal carriage at 1, 2, 6, 24, 36 and 48 weeks. | 1, 2, 6, 24, 36 and 48 weeks
  Decolonisation is determined by the following test outcomes:
  i. Negative PCR result (CP genes undetected) for stool sample subjected to direct PCR (Xpert Carba-R) ii. Negative PCR result (CP genes undetected) for stool sample subjected to culture on ChromID CARBA SMART media followed by PCR for suspected CPE colonies (Xpert Carba-R)
  At least one of the two tests have to be evaluable (clear positive or negative result obtained). Subject not meeting these criteria will be considered not-decolonised.
  If any one of the PCR results are positive, the subject is considered not-decolonised.
Progression to CPE infection | Up to 48 weeks
  Proportion of patients who progressed to CPE infection within 48 weeks, defined by isolation of CPE in a clinical isolate, compatible with an infective syndrome, as assessed by the study investigators.
Changes in stool microbiome | 1, 2, 6, 12, 24, 36, and 48 weeks
  Projected output from metagenomics analysis (i and ii) and culture-based assays (iii):
  i. Comparison of gut microbial composition at 1, 2, 6, 12, 24, 36, and 48 weeks after treatment with FMT or placebo with composition at pre-randomisation (including Shannon Diversity Index) ii. Comparison of relative abundance of CP producing and non-CP producing species at 1, 2, 6, 12, 24, 36, and 48 weeks after treatment with FMT versus placebo iii. CPE load in stool at 1, 2, 6, 12, 24, 36, and 48 weeks post-treatment
Frequency and severity of adverse events | Up to 48 weeks
  Comparison of the incidence and severity of all adverse events reported post-randomisation up to 48 weeks between the intervention and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Oon Tek Ng, MBBS, Principal Investigator — Tan Tock Seng Hospital

IPD SHARING:
Plan to Share IPD: No